CLINICAL TRIAL: NCT03209700
Title: Re-treatment for Partial or Non-responders for a Phase I Study of Autologous Mesenchymal Stromal Cell Coated Fistula Plug in Patients With Perianal Fistulas
Brief Title: Re-treatment From a Phase I Study of MSC-AFP in Patients With Perianal Fistulas
Acronym: MSC-AFP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: William A. Faubion, M.D. (Other)
Responsible Party: Sponsor-Investigator, William A. Faubion, M.D., William A. Faubion, M.D., Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-004503
Record Dates: First submitted 2017-07-03; First posted 2017-07-06 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Perianal Fistula; Cryptoglandular Perianal Fistula; Crohn's Perianal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MSC-AFP Single Treatment Group (Experimental): Eligible patients will be treated, single treatment group, no placebo arm
  Interventions: Drug: MSC-AFP

INTERVENTIONS:
Drug: MSC-AFP — Eligible patients will be treated with a fistula plug that has been coated with autologous mesenchymal stromal cells.
  Other Names: mesenchymal stromal cell coated fistula plug

SUMMARY:
This study is an extension to re-treat partial and non-responders from the previously approved Phase 1 MCS-AFP protocols IRB #12-009716 (Crohn's Disease perianal fistulas) and 15-003200 (cryptoglandular perianal fistulas).

DETAILED DESCRIPTION:
This study is an extension to re-treat partial and non-responders from the previously approved Phase 1 MCS-AFP protocols IRB #12-009716 (Crohn's Disease perianal fistulas) and 15-003200 (cryptoglandular perianal fistulas). This study will enroll patients that have persistent symptomatic perianal disease despite being treated with an MSC coated fistula plug, and also treat patients that have had recurrence of their perianal fistula.

As per the previously approval treatment under IND 15356, patients will have a single affected fistula treated, which is the same fistula that was treated in the original protocol. The matrix for delivering the cells is a Gore Bio-A Fistula Plug.

Subjects will be screened at outpatient clinic visits and interested qualified subjects will be offered participation in the trial and consented. At the first study visit (Visit 1; Screening visit), the patient will be evaluated and assessment will be made if an EUA is clinically necessary to assess the fistula. As this is a re-treatment trial, patients with incomplete response to initial plug placement typically have close follow up, recent MRI imaging, and may have a seton in place. If an EUA is clinically indicated, this would be by a colorectal surgeon for drainage of sepsis and placement of a seton as part of the standard clinical care for perianal fistula.

Patients will return on: Day 1, Week 4, Week 12, and Week 24.

ELIGIBILITY:
Inclusion Criteria

1. Males and females 18-65 years of age.
2. Residents of the United States.
3. Single draining perianal fistula for at least three months despite standard therapy
4. Concurrent therapies are permitted (such as antibiotics, corticosteroids, thiopurines).
5. Have no contraindications to MR evaluations: e.g. pacemaker or magnetically active metal fragments, claustrophobia
6. Ability to comply with protocol
7. Competent and able to provide written informed consent
8. Patients that were treated with an MSC-coated fistula plug in the study IRB#12-009716 or IRB#15-003200

Exclusion Criteria

1. Inability to give informed consent.
2. Clinically significant medical conditions within the six months before administration of MSCs: e.g. myocardial infarction, active angina, congestive heart failure or other conditions that would, in the opinion of the investigators, compromise the safety of the patient.
3. Specific exclusions: Evidence of hepatitis B, C, or HIV
4. History of cancer including melanoma (with the exception of localized skin cancers)
5. Investigational drug within thirty (30) days of baseline
6. A resident outside the United States
7. Previous allergic reaction to a perianal fistula plug.
8. Allergic to local anesthetics
9. Pregnant patients or trying to become pregnant or breast feeding.
10. Non-enterocutaneous tracts (i.e. recto-vaginal, entero-vesicular)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events (safety and toxicity). | 6-12 months
  Participants will have a health assessment and blood work measured at each study visit to monitor for adverse events, such as worsening of the perinal fistulizing disease, abnormal laboratory values, or significant abnormalities in physical examination. The Outcome Measure will be the number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment

SECONDARY OUTCOMES:
Number of participants with response to the treatment regarding potential cessation of drainage from their fistula. | 6 months
  Participants will have a clinical assessment of fistula drainage. Participants will be assessed during an office examination if their fistula is draining or not. The Outcome Measure will be the presence or absence of fistula drainage.

CONTACTS AND LOCATIONS:
Overall Officials: William A Faubion, M.D., Principal Investigator — Mayo Clinic; Eric J Dozois, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Minnesota, Rochester, Minnesota, United States